CLINICAL TRIAL: NCT04311242
Title: Microbiome Composition and Biomarker Discovery in Refractory Pediatric Epilepsy
Status: Withdrawn | Type: Observational
Why Stopped: Sponsor decision to not pursue epilepsy development.
Sponsor: Senda Biosciences (Industry)
Collaborators: Boston Children's Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: E-NEU-EPY-01
Record Dates: First submitted 2019-12-16; First posted 2020-03-17 (Actual); Last update posted 2021-02-26 (Actual); Status verified 2021-02

CONDITIONS: Epilepsy
MeSH Terms: conditions — Epilepsy | interventions — Diet

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Collecting blood and stool
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Diet — Ketogenic diet

SUMMARY:
Research study to look for bio markers in epilepsy patients on ketogenic diet

DETAILED DESCRIPTION:
Epilepsy is a neurological disorder characterized by the recurrence of unprovoked seizures that affects approximately 3.4 million people in the United States (1.2% of the total United States population) and more than 65 million people globally. The most commonly used treatments for epilepsy are antiepileptic drugs (AEDs); however, approximately 25% to 30% of the epilepsy population is considered pharmaco-resistant (characterized by the failure of ≥2 appropriately chosen and dosed AEDs).

Recent research suggests that the intestinal microbiota plays a central role in human health, and may play a role in a variety of central nervous system disorders, including seizure susceptibility. The microbiota has been shown to be associated with changes in factors relevant to neurotransmission, including neurotransmitter signaling, synaptic protein expression, long-term potentiation, and myelination. In addition to the microbiota's potential role in general neurotransmission, research suggests that the gut microbiome may differ between patients with pharmaco-resistant and pharmaco-sensitive epilepsies. Diet has been explored as an alternative form of therapy for patients with epilepsy, with the ketogenic diet showing promise as an alternative treatment for patients with drug-resistant epilepsy.

ELIGIBILITY:
Inclusion Criteria:

* Study participant and/or legal representative must be willing and able to give informed consent/assent for participation in the study.
* Study participant and/or legal representative must be willing and able to comply with all study requirements, in the opinion of the Investigator(s).
* Study participant is <18 years of age at the Screening Visit.
* Study participant has refractory epilepsy.

Exclusion Criteria:

* Study participant has a known cardiac disorder including arrhythmias or hypertension.
* Study participant has carnitine deficiency (primary), carnitine palmitoyltransferase I or II deficiency, or carnitine translocase deficiency.
* Study participant has beta-oxidation defects - medium-chain acyl dehydrogenase deficiency, long-chain acyl dehydrogenase deficiency, short-chain acyl dehydrogenase deficiency, long-chain 3-hydroxyacyl-coenzyme A deficiency, or medium-chain 3-hydroxyacyl-CoA deficiency.
* Study participant has a pyruvate carboxylase deficiency.
* Study participant has porphyria.
* Study participant is unable to maintain adequate nutrition.
* Study participant has a surgically remediable cause for refractory epilepsy.
* Study participant has a suspected mitochondrial disorder or has been diagnosed with a disorder in which a high-fat diet is contraindicated.
* Study participant has previously received a ketogenic diet or modified Atkins diet.
* Study participant has a chronic systemic disease like chronic kidney disease, chronic liver disease, heart disease (congenital and acquired), or chronic respiratory illness.
* Study participant's family is expected to have compliance problems with treatment and/or seizure registration.
* Study participant's seizures are under acceptable control.
* Study participant has had a vagus nerve stimulator implanted within the last 18 months, has started a new antiepileptic drug (AED) within the last 2 months, or has changed his/her antiepileptic drugs within the last month.
* Study participant has a medical condition, for example a metabolic disease, where ketogenic diet is contraindicated.
* Study participant's nutritional status is not good enough or intake of fluid is too small to permit treatment with ketogenic diet.
* Study participant has, within the last 2 months, been using medications or herbal medicine that have a considerable effect on glucose metabolism, such as oral glucocorticoids.
* Study participant has, within the last 2 months, been using medications or herbal medicine that have a considerable effect on metabolism of AEDs.
* Study participant uses herbal medicine which can interact with AEDs or a ketogenic diet.
* Study participant has participated in another study of an investigational drug within the previous 3 months before Screening (or within 5 half-lives for the investigational drug, whichever is longer) or is currently participating in another study of an investigational drug.

Ages: 1 Year to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: 50 epilepsy patients
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2020-04-15 (Actual); Primary Completion 2021-02-23 (Actual); Study Completion 2021-02-23 (Actual)

PRIMARY OUTCOMES:
Microbiome features associated with Ketogenic Diet response | 24 months
  Bacterial species and metabolomics biomarkers associated with patients responding to Ketogenic Diet

CONTACTS AND LOCATIONS:
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided